CLINICAL TRIAL: NCT03362268
Title: Efficacy and Safety of Intravenous IIaprazole for Peptic Ulcer Bleeding: A Randomized, Double-Blind, Omeprazole-Controlled, Multicenter, and Phase 2 Trail in China
Brief Title: IIaprazole for the Treatment and Prevention of Peptic Ulcer Bleeding in Chinese Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Livzon Pharmaceutical Group Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Livzon-IYI-Ⅱ
Record Dates: First submitted 2017-11-28; First posted 2017-12-05 (Actual); Last update posted 2017-12-06 (Actual); Status verified 2017-11

CONDITIONS: Peptic Ulcer Hemorrhage
MeSH Terms: conditions — Peptic Ulcer Hemorrhage | interventions — ilaprazole; Omeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ilaprazole (Experimental)
  Interventions: Drug: Ilaprazole
- omeprazole (Active Comparator)
  Interventions: Drug: omeprazole

INTERVENTIONS:
Drug: Ilaprazole — 10 mg ilaprazole daily (at day 1-3) through intravenous infusion within 30min with first dose doubling. Since 4th day, those patients were changed to take oral ilaprazole tablets 10mg each day till 30th day
  Arms: Ilaprazole
Drug: omeprazole — 40 mg omeprazole twice daily (at day 1-3) through intravenous infusion within 30min,Since 4th day, those patients were changed to take oral omeprazole tablets 20mg each day till 30th day
  Arms: omeprazole

SUMMARY:
The purpose of this study is to compare the efficacy and safety of ilaprazole and omeprazole in the treatment and prevention of peptic ulcer bleeding. Patients with endoscopically diagnosed peptic ulcer bleeding were enrolled in a randomized, double-blind, parallel and positive-controlled trial. They were randomly assigned into two groups, ilaprazole and omeprazole, to be treated for up to 30 days and be seen at day 3, 4, 7, 14 and 30. The primary endpoint was the hemostasis rate (hemostatic groups with endoscopy check ) and re-bleeding rate ( bleeding groups with endoscopy check) within 72 hours. Secondary end points include effective rate of hemostasis, mean volume of blood transfusion, the length of stay and re-bleeding rate, etc.

DETAILED DESCRIPTION:
Patients with endoscopically diagnosed gastric and duodenal ulcer bleeding were randomly assigned into two groups, ilaprazole and omeprazole. 120 patients were administrated 10 mg ilaprazole daily (at day 1-3) through intravenous infusion within 30min with first dose doubling. Since 4th day, those patients were changed to oral administration. Other 60 patients were administrated 40 mg omeprazole twice daily (at day 1-3) through intravenous infusion within 30min. Since 4th day, those patients were changed to oral administration. The efficacy of ilaprazole and omeprazole was evaluated by the primary endpoint including the hemostasis rate (hemostatic groups with endoscopy check ) and re-bleeding rate (bleeding groups with endoscopy check) within 72 hours and secondary end points including effective rate of hemostasis, average blood transfusion, the need to switch to other treatments (endoscopic treatment or surgery, etc.), hospital stay and re-bleeding rate at day 7, 14 and 30. Safety assessments based mainly on the occurrence, frequency, and severity of adverse events, which were monitored throughout the duration of the study, and also based on comprehensive indexes,including physical examination, electrocardiography, and routine laboratory investigations, which were performed at baseline and repeated at the end of the treatment period. For all adverse events, where necessary, patients were withdrawn from the study.This phase Ⅱ clinical trial was designed to compare the efficacy and safety of ilaprazole and omeprazole in the treatment and prevention of peptic ulcer bleeding.

ELIGIBILITY:
Inclusion Criteria:

1. were 18-65 years of age, male or female.
2. had symptoms of hematemesis, hematochezia, melena within 24 hours and clinically diagnosed as peptic ulcer bleeding.
3. had endoscopically diagnosed gastric or duodenal ulcer bleeding (multiple ulcers was judged by the higher Forrest level).
4. were patients of Forrest Ⅰa-Ⅱb level and had successful endoscopic surgery to stop bleeding (bleeding was cured and the blood vessels were flat or became into the lumen). Ⅱc-Ⅲ grade patients did not receive endoscopic hemostasis.
5. voluntarily sign informed consent.

Exclusion Criteria:

1. had hemorrhagic shock (systolic blood pressure<90mmHg) or require surgery.
2. were non-ulcer bleeding and gastric ulcer biopsy proved malignant.
3. had gastrectomy and gastrointestinal anastomosis.
4. were suffering from serious heart, liver, brain, lung, kidney and other serious diseases.
5. had coagulation disorders (laboratory tests showed that platelets <80 × 109 / L, PT abnormal and exceed the normal control for 3 seconds, APTT than the normal control for 10 seconds).
6. had hypersensitivity or idiosyncratic reaction to ilaprazole, omeprazole, esomeprazole or any other benzimidazole.
7. had positive result of urine pregnancy test.
8. used the same kind of drugs within 48 hours before entering the group.
9. need to continue the combination of the following drugs that have an effect on treatment during the study: NSAIDs, corticosteroids, heparin, warfarin and vitamin K, platelet antagonists or other hemostatic agents.
10. participated in a clinical trial with an investigational drug or device within the past three months.
11. had alcoholic intemperance, drug addiction or other factors that researchers think it unfit for drug clinical trials.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
The rate of hemostasis peptic ulcer hemorrhage patients | 72 hours
  Measure: The hemostasis rate checked by endoscopy within 72 hours